CLINICAL TRIAL: NCT00998374
Title: Comparison Between Pyloric Preserving and Non-Pyloric Preserving Bariatric Surgery With Glucose Challenge
Status: Completed | Type: Observational
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Other Study IDs: AS08018
Record Dates: First submitted 2009-10-15; First posted 2009-10-20 (Estimated); Results first posted 2014-04-21 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-03

CONDITIONS: Hypoglycemia; Obesity
MeSH Terms: conditions — Hypoglycemia; Obesity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pyloric-sparing vs. non-pyloric sparing: Pyloric: SG & DS Non-pyloric: RYGB

SUMMARY:
This study will compare glucose and simple carbohydrate sensitivity. The hypothesis is that rapid emptying of high-glycemic index foods after Roux-En-Y gastric bypass (RYGB) causes reactive hypoglycemia. It is believed that the controlled release offered by an intact pylorus will be advantageous for long term results in bariatric surgery. This study can provide a scientific rationale, in a short duration of time, for why pylorus sparing surgery, such as the sleeve gastrectomy or duodenal switch, may offer therapeutic advantages, as compared to non-pyloric sparing surgery, namely the gastric bypass.

DETAILED DESCRIPTION:
Clinical Trial Objective:

The objective of this clinical trial is to determine whether an intact pylorus prevents reactive hypoglycemia following challenge with liquid glucose preparation and/or solid load made of refined flour product that is a simple carbohydrate.

Clinical Trial Design:

This is a prospective, non-randomized, clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* The patient is greater than 18 years old;
* The patient has a BMI > 35;
* Patient meets standards for bariatric surgery;

Exclusion Criteria:

* The patient has an incurable malignant or debilitating disease;
* The patient has been diagnosed with a severe eating disorder;
* The patient is currently pregnant (pregnancy test required for confirmation for those of child bearing years);
* The patient is unable to comply with the study requirements, follow-up schedule, or to give valid informed consent

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients >18 years of age BMI greater than or equal to 35
Sampling Method: Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2009-09; Primary Completion 2013-01 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Roslin, MD, Principal Investigator — Lenox Hill Hospital
Locations (1):
- Lenox Hill Hospital 186 E76th Street, 1st Floor, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Pyloric-sparing: Pyloric: Sleeve Gastrectomy (SG) & Duodenal Switch (DS)
- Non-pyloric Sparing: Non-pyloric sparing: Roux-en-Y Gastric Bypass (RYGB)
Period: Overall Study
Arm/Group | Pyloric-sparing | Non-pyloric Sparing
Started | 39 | 23
Completed | 27 | 12
Not Completed | 12 | 11

BASELINE CHARACTERISTICS:
Groups:
- Pyloric-sparing: Pyloric sparing: Sleeve Gastrectomy and Duodenal Switch
- Non-pyloric Sparing: Non-pyloric sparing: Roux-en-Y Gastric Bypass
- Total: Total of all reporting groups
Arm/Group | Pyloric-sparing | Non-pyloric Sparing | Total
Number analyzed (Participants) | 39 | 23 | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 39 | 23 | 62
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 20 | 44
  Male | 15 | 3 | 18
Region of Enrollment [Number; unit: participants]
  United States | 39 | 23 | 62

OUTCOME MEASURES:

1. Primary Outcome: Mean Serum Glucose Levels
Description: Serum glucose levels measured to assess reactive hypoglycemia status
Time Frame: 30, 60, and 120 minutes at 6, 9, and 12 months post-operatively
Measure: Mean (Standard Deviation); unit: mg/dl
Groups:
- Pyloric-sparing: Pyloric: SG & DS
- Non-pyloric Sparing: Non-pyloric sparing: RYGB
Arm/Group | Pyloric-sparing | Non-pyloric Sparing
Number analyzed (Participants) | 39 | 23
mg/dl
  6 months - 30 minutes | 123.1 (48.8) | 157.5 (56.2)
  9 months - 30 minutes | 103.2 (30.2) | 138 (50.1)
  12 months - 30 minutes | 130.3 (49.6) | 173.4 (78.3)
  6 months - 60 minutes | 121.8 (65.6) | 152.6 (79.6)
  9 months - 60 minutes | 98.8 (34.9) | 132.6 (65.2)
  12 months - 60 minutes | 121.1 (52.3) | 141.8 (90.7)
  6 months - 120 minutes | 83.4 (48.4) | 83.4 (45.9)
  9 months - 120 minutes | 88.3 (33.1) | 85.3 (41.3)
  12 months - 120 minutes | 84.5 (52.1) | 79.5 (58.6)

2. Secondary Outcome: Insulin Resistance
Description: Measured by levels of post prandial insulin
Time Frame: 6, 9, and 12 months post-operatively
Measure: Mean (Standard Deviation); unit: pmol/L
Groups:
- Non-pyloric Sparing: Non-pyloric: RYGB
Arm/Group | Pyloric-sparing | Non-pyloric Sparing
Number analyzed (Participants) | 39 | 23
pmol/L
  1 hour pp - 6 month | 13.7 (11.7) | 21.2 (16.4)
  1 hour pp - 9 month | 6.4 (3.2) | 20.9 (25.1)
  1 hour pp - 12 month | 10.9 (9.3) | 16.7 (14.6)
  2 hours pp - 6 month | 3.8 (2.5) | 3.9 (6.7)
  2 hours pp - 9 month | 2.6 (2.3) | 4.2 (4.9)
  2 hours pp - 12 month | 4.8 (12.4) | 6.6 (12.3)

3. Secondary Outcome: Subjective Symptoms of Hypoglycemia During Glucose Tolerance Testing
Description: Subjective symptoms of hypoglycemia during glucose tolerance testing measured by patients' responses to a questionnaire about symptoms of Weakness, Nausea, Hunger, Headache, Dizziness, Diaphoresis graded on a yes/no response
Time Frame: 6, 9, and 12 months post-op
Measure: Number; unit: participants
Groups:
- Non-pyloric: Non-pyloric: RYGB
Arm/Group | Pyloric-sparing | Non-pyloric
Number analyzed (Participants) | 39 | 23
participants
  6 Month - Weakness | 6 | 8
  9 Month - Weakness | 1 | 3
  12 Month - Weakness | 2 | 6
  6 Month - Nausea | 12 | 8
  9 Month - Nausea | 2 | 6
  12 Month - Nausea | 5 | 6
  6 Month - Hunger | 4 | 3
  9 Month - Hunger | 0 | 2
  12 Month - Hunger | 2 | 1
  6 Month - Headache | 4 | 3
  9 Month - Headache | 3 | 3
  12 Month - Headache | 4 | 3
  6 Month - Dizziness | 10 | 7
  9 Month - Dizziness | 1 | 4
  12 Month - Dizziness | 0 | 3
  6 Month - Sweating | 4 | 2
  9 Month - Sweating | 0 | 2
  12 Month - Sweating | 0 | 2

4. Primary Outcome: Reactive Hypoglycemia Status
Description: Postoperative reactive hypoglycemia was defined as either
  * serum glucose <60 mg/dL at least 1 hour after initiation of glucose tolerance testing
  * serum glucose decrease ≥100 mg/dL within 1 hour after initiation of glucose tolerance testing
Time Frame: 6 months, 9 months, 12 months post-op
Measure: Number; unit: participants
Arm/Group | Pyloric-sparing | Non-pyloric Sparing
Number analyzed (Participants) | 39 | 23
participants
  6 Month | 11 | 6
  9 Month | 4 | 3
  12 Month | 7 | 7

ADVERSE EVENTS:
Time Frame: Day 0, 2 weeks, 4 weeks, 3 months, 6 months, 9 months, 12 months
Description: During each visit study subjects were asked whether an adverse event had occurred, and their 'yes'/'no'responses were recorded on the corresponding visit CRFs.
Arm/Group | Pyloric-sparing | Non-pyloric Sparing
Serious Adverse Events (participants affected / at risk) | 5/39 | 3/23
Other Adverse Events (participants affected / at risk) | 8/39 | 2/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pyloric-sparing (N=39) | Non-pyloric Sparing (N=23)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anastamotic Leak (Surgical and medical procedures) | 1 (1) | 0 (0)
DVT/PE (Vascular disorders) | 1 (1) | 0 (0)
Lower Left Quadrant (LLQ) pain (General disorders) | 1 (1) | 0 (0)
Portal and superior mesenteric venous thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Epigastric hernia (General disorders) | 1 (1) | 0 (0)
Hypoalbuminemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Bleeding (Surgical and medical procedures) | 0 (0) | 1 (1)
Enterocutaneous fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pyloric-sparing (N=39) | Non-pyloric Sparing (N=23)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0)
Hypovolemia (General disorders) | 1 (1) | 0 (0)
Hypoxic (General disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Left Kidney Stone (left flank pain) (General disorders) | 1 (1) | 0 (0)
more than expected post-op pain (General disorders) | 1 (1) | 0 (0)
Nocturnal desaturation (General disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
SVT (Cardiac disorders) | 1 (1) | 0 (0)
Anastomotic stricture (Surgical and medical procedures) | 1 (1) | 0 (0)
GERD (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mild tingling of the legs (General disorders) | 1 (1) | 0 (0)
Incomplete staple line (Surgical and medical procedures) | 0 (0) | 1 (1)
Severe vomiting (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No